CLINICAL TRIAL: NCT04846179
Title: To Evaluate the Effect of Ginkgo Biloba Extract on Optic Nerve Head Perfusion
Brief Title: To Evaluate the Effect of Ginkgo Biloba Extract on Optic Nerve Head Perfusion Examined Using OCTA
Acronym: GBE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1026588
Record Dates: First submitted 2021-04-12; First posted 2021-04-15 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Glaucoma
Keywords: Ginkgo biloba extract; Ocular perfusion; Optical coherence tomography angiography
MeSH Terms: conditions — Glaucoma | interventions — Ginkgo biloba extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ginkgo biloba extract group (Experimental): Group receiving ginkgo biloba extract supplementation
  Interventions: Dietary Supplement: Ginkgo biloba extract

INTERVENTIONS:
Dietary Supplement: Ginkgo biloba extract — Patients recruited to Ginkgo Biloba Extract (GBE) group will be advised to take Webber Natural Ginkgo Biloba 120 mg soft gel, 1 tablet twice a day for 4 months.

SUMMARY:
Glaucoma is defined as progressive neuropathy of the optic nerve. It is an important cause of irreversible blindness worldwide. Lowering the intraocular pressure is the only proven treatment for this neurodegenerative disease. However, there is ongoing research looking at another modifiable risk factor that affects the development and progression of this disease. Ginkgo biloba (Ginkgoacease) is a tree species that has been used in traditional medicine for several hundred years to treat various diseases include improving vascular perfusion. We propose a study examining the effect of Ginkgo biloba extract supplementation on ocular perfusion using optical coherence tomography angiography.

DETAILED DESCRIPTION:
Glaucoma is defined as progressive neuropathy of the optic nerve. It is an important cause of irreversible blindness worldwide. Lowering the intraocular pressure is the only proven treatment for this neurodegenerative disease. However, there is ongoing research looking at another modifiable risk factor that affects the development and progression of this disease. There is growing evidence that vascular dysfunction plays a role in the pathogenesis of glaucoma. Low ocular perfusion pressure (OPP), which is expressed as the difference between mean arterial pressure and intraocular pressure (IOP), has been hypothesized to lead to glaucomatous optic neuropathy via ischemic damage to the optic nerve. The Barbados Eye Study showed that reduced OPP at baseline was associated with a three-fold increased risk of glaucoma development. Evidence has also shown that optic nerve hypoperfusion may contribute to the progression of glaucoma.

Ginkgo biloba (Ginkgoacease) is a tree species that has been used in traditional medicine for several hundred years to treat various diseases. There have been recent studies that have examined its medicinal properties in treating age-related cognitive disease and neuronal degeneration resulting from ischaemic events. Studies examining systemic vascular ischemic diseases have shown a beneficial effect of ginkgo Biloba extract (GBE) on systemic arterial occlusive diseases. There is also preliminary research examining the effect GBE has on optic nerve head perfusion in patients with glaucoma. There is a study that examined the effects of antioxidants including GBE on ocular blood flow in patients with glaucoma using doppler ultrasound. When compared with patients receiving placebo, patients after antioxidant therapy containing GBE were shown to have increased peak systolic and/or end-diastolic blood velocities in all retrobulbar blood vessels, reduced vascular resistance in the central retinal and nasal short posterior ciliary arteries, increased superior and inferior temporal retinal capillary mean blood flow, an increased ratio of active to nonactive retinal capillaries. In the area of optic nerve head perfusion studies, fluorescein angiography has also been used in investigating alteration in blood flow in glaucomatous versus normal eyes. However, utility in clinical practice is limited by the qualitative nature of the test and the risk for adverse events. While color Doppler ultrasound is greatly limited in terms of resolution and can be openly used to examine large vessels of the eye. New development in ocular imaging has shown that OCTA can provide reproducible and quantifiable information about the microvasculature of the optic nerve and peripapillary retina in patients with glaucoma and can do so in a rapid and non-invasive manner avoiding some of the limitations on doppler ultrasound and fluorescein angiography.

GBE Egb761 is a standardized GBE that's used in most published research on the effect of ginkgo Biloba. It is a standardized GBE used in evidence-based medicine and clinical investigations ensuring clinical standardization and a safe manufacturing process. It has much of the toxic ginkgolic acid removed leaving behind the active components of flavonoid glycosides and terpene lactones. In general, GBE is well tolerated with a low side effect profile. Several systematic reviews on research using GBE (daily dose of up to 600 mg) report no statistical difference in side effects with GBE compared with placebo. There have been some concerns regarding the bleeding risk while on ginkgo supplementation. However, randomized placebo-controlled studies in healthy volunteers have not shown any changes in bleeding time, coagulation parameters, or platelet function. Multiple studies have reported minimal adverse effects (AEs) of GBE within a specific prescribed dosage range. Overall, GBE continues to be a well-tolerated supplement with a low side effect profile. Systematic reviews of the Cochrane databases, PubMed/MEDLINE, EMBASE, and Google Scholar, report no statistically significant difference in AEs between 80 and 600 mg of GBE and placebo.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Early open angle glaucoma based on gonioscopy, clinical assessment of optic nerve head, OCT optic nerve and Humphrey Visual Field 24-2 (MD < -10dB) and positive Glaucoma Hemifield Test
* BCVA equal or better than 6/12
* Written consent
* Ability to comply with treatment intervention for duration of study

Exclusion Criteria:

* Younger than 18 years of age
* Angle closure glaucoma or secondary open angle glaucoma
* Refraction exceeding 6D spherical equivalent or 3D astigmatism
* Severe corneal, lens, vitreous media opacity limit signal strength of OCTA imaging
* Severe open angle glaucoma with visual field mean deviation worse than -10dB
* Inability to comply to treatment intervention (e.g. swallowing difficulty)
* History of ocular disease affecting ocular perfusion (e.g. CRAO, CRVO, diabetic retinopathy, ocular ischemic syndrome, ischemic optic neuropathy)
* History of glaucoma surgery
* Those taking anticoagulant therapy
* Those with blood disorders or diabetes
* Women who were pregnant, planning to become pregnant, or who were breast-feeding,
* Patients with a history of seizures or who were currently taking anti-convulsant medication, and
* Taking any drugs that may interact with GBE

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Optic nerve head and macula perfusion | 4 months
  Optic nerve head and macula perfusion will be analyzed using optical coherence tomography angiography after 4 months of ginkgo biloba extract supplementation

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Scotia Health, Halifax, Nova Scotia, Canada